CLINICAL TRIAL: NCT01708317
Title: The Use of Computer-Assisted Self-Interviews to Improve Adolescent and Young Adult Health Screening in the Pediatric Emergency Department
Brief Title: Computer-Assisted Self-Interviews and Health Screening in the Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: St. Louis Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20110243
Record Dates: First submitted 2012-10-09; First posted 2012-10-16 (Estimated); Results first posted 2013-01-08 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2012-12

CONDITIONS: Gonorrhea; Chlamydia
Keywords: ACASI; Gonorrhea; Chlamydia; Emergency Department; Youth; Adolescents; Computer; Questionnaire
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACASI (Other): The group of patients that agreed to participate in the study and answer questions on our Audio-enhanced Computer-Assisted Self-Interview (ACASI)
  Interventions: Behavioral: ACASI

INTERVENTIONS:
Behavioral: ACASI — Youth who participated in this study completed the ACASI -- they provided details about their sexual history, and the software program used their responses to create a recommendation for chlamydia/gonorrhea testing. The information obtained through the ACASI was integrated into the emergency department (ED) electronic medical record. ED physicians and nurses were able to review the information and order chlamydia/gonorrhea testing if needed.

SUMMARY:
The purpose of this study is to determine if an Audio-enhanced Computer-Assisted Self-Interview (ACASI) will lead to increase testing for sexually transmitted infections in youth visiting a pediatric ED

DETAILED DESCRIPTION:
The purpose of this study is to see if computer based health surveys for teenagers and young adults in the emergency department can improve the care we give, even for things that are not related to why they came to the emergency department.

Topics that are important in this age range include depression, violence, sexual behavior, physical activity and nutrition, though we are not asking about all of these.

WHAT WILL HAPPEN DURING THIS STUDY?

We wish to respect the privacy of everyone takes this survey. In order to do this, we are asking all relatives including your parents or guardians to respect several things so that you may participate:

* We cannot tell family or friends the exact questions on the survey
* You must be given complete privacy to answer the questions
* The answers will only be shown to the healthcare team taking care of them today and the people running the study - family members will not be shown the answers
* Family and friends will not pressure you to discuss the survey or their answers after you are done
* You will be given privacy to discuss their answers with the healthcare team

If you do not feel your friends and family can respect these requests, then you cannot take the survey and cannot enroll in the study.

If you agree to these requests, we will use a private area and allow you to use a computer to do the following:

* Explain in more detail what types of questions we will ask and why they are important
* Tell you how we will use your answers to improve their health care
* Give you a chance to answer any questions you have about the study
* Answer a series of questions about yourself and your health

You are allowed to skip any questions you do not want to answer and can stop at any time.

After you have completed the survey, a summary of your answers will become part of your medical record from today and be shown to the doctors and nurses taking care of you today.

Most participants will be asked to review their answers in private with the doctors and nurses taking care of them. If you do, your family and friends will be asked to step out of the room while you review the answers with the doctors and nurses.

Some participants may have additional testing or services done as part of their visit today based on their answers

ELIGIBILITY:
Inclusion Criteria:

* Patient in the St. Louis Children's Hospital Emergency Department
* 15-21 years old

Exclusion Criteria:

* Evaluation of abuse or sexual assault
* Activation of the trauma system,
* Level 1 or 2 triage scores (highest severity)
* Disabilities preventing independent computer use
* Psychiatric chief complaints
* Inability to speak English

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 801 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fahd A Ahmad, MD, MSCI, Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Porter SC, Silvia MT, Fleisher GR, Kohane IS, Homer CJ, Mandl KD. Parents as direct contributors to the medical record: validation of their electronic input. Ann Emerg Med. 2000 Apr;35(4):346-52. doi: 10.1016/s0196-0644(00)70052-7. PMID 10736120
- [Background] Bachman JW. The patient-computer interview: a neglected tool that can aid the clinician. Mayo Clin Proc. 2003 Jan;78(1):67-78. doi: 10.4065/78.1.67. PMID 12528879
- [Background] Porter SC, Mandl KD. Data quality and the electronic medical record: a role for direct parental data entry. Proc AMIA Symp. 1999:354-8. PMID 10566380
- [Background] Porter SC, Cai Z, Gribbons W, Goldmann DA, Kohane IS. The asthma kiosk: a patient-centered technology for collaborative decision support in the emergency department. J Am Med Inform Assoc. 2004 Nov-Dec;11(6):458-67. doi: 10.1197/jamia.M1569. Epub 2004 Aug 6. PMID 15298999
- [Background] Williams ML, Freeman RC, Bowen AM, Zhao Z, Elwood WN, Gordon C, Young P, Rusek R, Signes CA. A comparison of the reliability of self-reported drug use and sexual behaviors using computer-assisted versus face-to-face interviewing. AIDS Educ Prev. 2000 Jun;12(3):199-213. PMID 10926124
- [Background] Kissinger P, Rice J, Farley T, Trim S, Jewitt K, Margavio V, Martin DH. Application of computer-assisted interviews to sexual behavior research. Am J Epidemiol. 1999 May 15;149(10):950-4. doi: 10.1093/oxfordjournals.aje.a009739. PMID 10342804
- [Background] Millstein SG, Irwin CE Jr. Acceptability of computer-acquired sexual histories in adolescent girls. J Pediatr. 1983 Nov;103(5):815-9. doi: 10.1016/s0022-3476(83)80493-4. PMID 6631616
- [Background] Hewett PC, Mensch BS, Erulkar AS. Consistency in the reporting of sexual behaviour by adolescent girls in Kenya: a comparison of interviewing methods. Sex Transm Infect. 2004 Dec;80 Suppl 2(Suppl 2):ii43-8. doi: 10.1136/sti.2004.013250. PMID 15572639

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We monitored overall testing in the ED from Jan 2010 - March 2012, but only actively enrolled patients from April 18, 2011 - Dec 20, 2011. All ACASI participants were patients in the St. Louis Children's Hospital ER.
Pre-assignment Details: There was an education lead in before introducing the ACASI, to see if education alone would increase the amount of patients receiving gonorrhea/chlamydia testing. The education started in Jan, 2011 and continued the remainder of the study period.
Groups:
- ACASI: The group of patients that agreed to participate in the study and answer questions on our Audio-enhanced Computer-Assisted Self-Interview (ACASI)
  ACASI : Youth who participated in this study completed the ACASI -- they provided details about their sexual history, and the software program used their responses to create a recommendation for chlamydia/gonorrhea testing. The information obtained through the ACASI was integrated into the emergency department (ED) electronic medical record. ED physicians and nurses were able to review the information and order chlamydia/gonorrhea testing if needed.
  We compared testing over 4 time periods: 2010 (baseline), Jan - April 17, 2011 (education only), April 18-2011 - Dec 20, 2011 (education + enrollment in ACASI), and Dec 21, 2011 - March 31, 2012 (education only, ACASI enrollment stopped.
Period: 2010 Control Period
Arm/Group | ACASI
Started | 3929 (# of ED patients eligible for ACASI, had it been available, in control period)
Completed | 3929
Not Completed | 0
Period: Initial Education Period
Arm/Group | ACASI
Started | 982 (# of ED patients eligible for ACASI, had it been available, in initial education period)
Completed | 982
Not Completed | 0
Period: ACASI + Education Period
Arm/Group | ACASI
Started | 2601 (# of ED patients eligible for ACASI in the period the ACASI was actually available.)
Completed | 2601
Not Completed | 0
Period: Final Education Period
Arm/Group | ACASI
Started | 909 (# of ED patients eligible for ACASI, had it been available, in final education period)
Completed | 909
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ACASI
Number analyzed (Participants) | 8421
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7042
  Between 18 and 65 years | 1379
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 17.0 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4643
  Male | 3778
Region of Enrollment [Number; unit: participants]
  United States | 8421

OUTCOME MEASURES:

1. Primary Outcome: Gonorrhea and Chlamydia Testing in the Pediatric ED
Description: The primary outcome was change in the proportion of adolescent patients receiving chlamydia and gonorrhea testing rates during their ED visit over 4 time periods.
  Period 1) 2010 testing as a historical control Period 2) Jan 2011, began providing staff education about the risks of gonorrhea/chlamydia and need for increased testing Period 3) Education continues, but enrolled patients in the ACASI from April 18, 2011 - Dec 20, 2011.
  Period 4) ACASI enrollment completed, education continued through March 2012
  We specifically analyzed gonorrhea/chlamydia testing among ED patients that would have been eligible to take the ACASI, had it been continuously available throughout these time periods. We did this to isolate the effects on testing by the ACASI vs. education alone.
Time Frame: 27 months
Population: We analyzed every patient in this time period that met our ACASI inclusion/exclusion criteria
Measure: Number; unit: percentage of participants
Groups:
- Historical Control: Participants seen in SLCH ED in 2010 that met ACASI inclusion/exclusion criteria
- Initial Education Period: Participants seen in SLCH ED Jan 1 - April 17 2011 during initial education period that met ACASI inclusion/exclusion criteria
- ACASI + Education: Participants seen in SLCH ED April 18 - Dec 20 2011 that met ACASI inclusion/exclusion criteria. During this period education continued and ACASI enrollment was conducted.
- Final Education Period: Participants seen in SLCH ED Dec 21, 2011 through March 2012 that met ACASI inclusion/exclusion criteria. During this period education continued and no ACASI enrollment was conducted.
Arm/Group | Historical Control | Initial Education Period | ACASI + Education | Final Education Period
Number analyzed (Participants) | 3929 | 982 | 2601 | 909
percentage of participants | 9.7 | 9.3 | 17.8 | 12.4
Statistical Analysis 1: Comparison: Historical Control vs Initial Education Period vs ACASI + Education vs Final Education Period; We compared testing in the 4 time frames described, including the time frame in which we enrolled patients in the ACASI; Test type: Superiority or Other; p < .001, Chi-squared — We used a cutoff of P<0.05 as statistically significant; 3 degrees of freedom to compare 4 time periods; Mean Difference (Final Values) = 5

ADVERSE EVENTS:
Time Frame: April 18, 2011 - Dec 20, 2011
Description: This is the time frame in which ACASI enrollment occurred
Arm/Group | ACASI
Serious Adverse Events (participants affected / at risk) | 0/801
Other Adverse Events (participants affected / at risk) | 0/801

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No